CLINICAL TRIAL: NCT01222416
Title: Positron Emission Tomography (PET)-Computed Tomography (CT) PET/CT Evaluation of Treatment Response in Breast Cancer
Brief Title: PET/CT Evaluation of Treatment Response in Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Associate Professor; Radiation Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC BRE 09108
Record Dates: First submitted 2010-09-29; First posted 2010-10-18 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorodeoxyglucose F18; Radiopharmaceuticals; alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fluorodeoxyglucose PET/CT (FDG-PET/CT) (Experimental): A PET/CT scan prior to the initiation of therapy, and then two additional scans following the initiation of therapy. Each patient will have up to three scans in a 6 month time frame.
  Interventions: Radiation: Radiopharmaceutical Administration [18F]-FDG
- fluorodeoxythymidine PET/CT (FLT-PET/CT) (Experimental): A PET/CT scan prior to the initiation of therapy, and then two additional scans following the initiation of therapy. Each patient will have up to three scans in a 6 month time frame.
  Interventions: Radiation: Radiopharmaceutical: [18F]-FLT

INTERVENTIONS:
Radiation: Radiopharmaceutical Administration [18F]-FDG — Adult dose: (0.15 mCi/kg ranging from 3 to 16 mCi,route IV. Time interval between administration and scanning: 60 +/- 10minutes post-injection.
  Arms: fluorodeoxyglucose PET/CT (FDG-PET/CT)
Radiation: Radiopharmaceutical: [18F]-FLT — Adult dose: (0.15 mCi/kg ranging from 3 to 16 mCi), route = IV, Time interval between administration and scanning: 60 +/- 10minutes post-injection.
  Arms: fluorodeoxythymidine PET/CT (FLT-PET/CT)

SUMMARY:
The purpose of this study is to develop Positron Emission Tomography (PET) - Computed Tomography (CT) PET/CT imaging methods for looking at the effects of chemotherapy in breast cancer.

ELIGIBILITY:
Inclusion Criteria

* Subjects must have histologically proven breast cancer
* Subjects are being considered for preoperative chemotherapy
* Subjects must be ≥ 18 years old. Sensor Sub-Study Only
* Palpable subcutaneous or known disease with one surface <1cm below surface of skin.
* A subset of patients who have a mass located on any surface of the breast that is accessible for Lucerno sensor placement will have additional testing.

Exclusion Criteria

* Children will be excluded from this study.
* Pregnant women and women who are breast feeding will be excluded from this study. (The Vanderbilt University Medical Center radiology "PET Procedure Screening Form" will be used to identify and exclude subjects who are pregnant or breastfeeding. A urine pregnancy test/or serum beta HCG will also be performed for women of child bearing potential).
* Patients who are acutely ill who are deemed by their treating physician as not suitable candidates for this study.
* Intraluminal lesions will be excluded from the sensor sub-study.
* Non biopsy proven malignancy will be excluded from this study.
* Palpable subcutaneous or known disease with one surface >1cm below surface of skin will be excluded from the sensor sub-study.
* Draining or exposed malignant tumor will be excluded from the sensor sub-study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial opened to accrual on 10/13/2010 and closed to accrual on 4/14/2015.
Pre-assignment Details: No participants were enrolled onto the Fluorodeoxythymidine PET/CT (FLT-PET/CT) arm because this trial closed to accrual early due to slow accrual.
Period: Overall Study
Arm/Group | Fluorodeoxyglucose PET/CT (FDG-PET/CT) | Fluorodeoxythymidine PET/CT (FLT-PET/CT)
Started | 50 | 0
Completed | 30 | 0
Not Completed | 20 | 0
Not completed — ineligible;metastasis | 3 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — scheduling | 6 | 0
Not completed — missed view/scan | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects must have histologically proven breast cancer
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluorodeoxyglucose PET/CT (FDG-PET/CT) | Fluorodeoxythymidine PET/CT (FLT-PET/CT) | Total
Number analyzed (Participants) | 50 | 0 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 |  | 46
  >=65 years | 4 |  | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 |  | 50
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 |  | 2
  Not Hispanic or Latino | 48 |  | 48
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 |  | 1
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 11 |  | 11
  White | 37 |  | 37
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 |  | 50

OUTCOME MEASURES:

1. Primary Outcome: The Difference in the Change (Pre and End-treatment) of Standard Uptake Value (SUV) Between Pathological Non-responders and Responders (pCR)
Description: The quantitative measures of standard uptake value (SULpeak and SULmax, prone and supine position) from PET were obtained. SUV = (Tracer activity in tissue)/(Injected radiotracer dose/patient weight or lean body mass) with unit microcuries/g/(millicuries/kg) (no unit after simplification). The SUV was averaged over the tumor regions. These averages were computed for each patient at each time point. All patients were were planned to be scanned three times: prior to treatment, during treatment and at the end of treatment. The change of SUV was calculated as the end of treatment value minus the pre-treatment value. Then the difference in the change between the responders and non-responders were estimated using Wilcoxon rank sum test. The pseudomedians and nonparametric confidence intervals for the difference (change of non-responders minus the change of responders) were reported for parameters SULpeak and SULmax measured for different positions. Pathological response were measured at the
Time Frame: up to 6 months (1 scan prior to chemotherapy and 2 scans prior to surgery)
Population: 19 Patients had the scanned data at two time points: prior treatment and at the end of treatment.
Measure: Median (95% Confidence Interval); unit: microcuries/g/(millicuries/kg)
Arm/Group | Fluorodeoxyglucose PET/CT (FDG-PET/CT) | Fluorodeoxythymidine PET/CT (FLT-PET/CT)
Number analyzed (Participants) | 19 | 0
microcuries/g/(millicuries/kg)
  Difference in SULpeak change, prone | 1.23 [-2.01 to 3.82] |
  Difference in SULmax change, prone | 2.12 [-1.87 to 4.45] |
  Difference in SULpeak change, supine | 1.89 [-1.37 to 4.70] |
  Difference in SULmax change, supine | 2.88 [-1.53 to 5.93] |

2. Secondary Outcome: Compare and Combine Magnetic Resonance Imaging (MRIs) (Obtained From Study BRE0588) and Positron Emission Tomography/ Computed Tomography (PET/CT) Methods to Develop a Robust Assessment of Tumor Status.
Time Frame: 48 months
Population: There were insufficient number of patients who had both MRI and PET performed to allow for meaningful statistical comparisons.
Arm/Group | Fluorodeoxyglucose PET/CT (FDG-PET/CT) | Fluorodeoxythymidine PET/CT (FLT-PET/CT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Study personnel are responsible for the accurate documentation, investigation and follow-up of all adverse events and unanticipated problems involving risks to participants and others that are possibly related to study participation.
Arm/Group | Fluorodeoxyglucose PET/CT (FDG-PET/CT) | Fluorodeoxythymidine PET/CT (FLT-PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/0
Other Adverse Events (participants affected / at risk) | 0/50 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes